CLINICAL TRIAL: NCT04579393
Title: A Phase II Study Evaluating Fostamatinib for Hospitalized Adults With COVID-19
Brief Title: Fostamatinib for Hospitalized Adults With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10000110; 000110-H
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-05

CONDITIONS: Coronavirus Disease 2019
Keywords: SARS-CoV-2; Cytokines; Spleen Tyrosine Kinase; ARDS
MeSH Terms: conditions — COVID-19 | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): fostamatinib in combination with standard of care (SOC) for the treatment of COVID-19
  Interventions: Drug: fostamatinib
- Intervention - Placebo (Placebo Comparator): Placebo in combination with standard of care (SOC) for the treatment of COVID-19
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo tablets to match fostamatinib 100 mg and 150 mg will be provided.
  Arms: Intervention - Placebo
Drug: fostamatinib — The study intervention is fostamatinib, an inhibitor of spleen tyrosine kinase that will be administered orally at a dose of 150 mg twice daily for 14 days or 28 doses. Subjects will receive standard of care and be randomized to receive fostamatinib or matching placebo.
  Arms: Intervention

SUMMARY:
Background:

COVID-19 is a new disease caused by SARS-CoV-2 that was identified in 2019. Some people who get sick with COVID-19 become ill requiring hospitalization. There are some medicines that may help with recovery. Researchers want to see if a drug called fostamatinib may help people who are hospitalized with COVID-19.

Objective:

To learn if fostamatinib is safe in patients who are hospitalized with COVID-19 and gain earlier insight into whether it improves outcomes.

Eligibility:

Adults age 18 and older who are hospitalized with COVID-19.

Design:

Participants will be screened with a physical exam, including vital signs and weight. They will have a blood test and chest x-ray. They will have a COVID-19 test as a swab of either the back of the throat or the back of the nose. They will take a pregnancy test if needed.

Participants will be randomly assigned, to take either fostamatinib pills or a placebo twice daily for up to 14 days in addition to standard of care for COVID-19. If they can swallow, they will take the pills by mouth with water. If they cannot swallow or are on mechanical ventilation, the pills will be crushed, mixed with water, and given through a tube placed through the nostril, or placed in the mouth, down the esophagus, and into the stomach. Blood samples will be taken daily. Participants will return to the Clinical Center for safety follow-up visits. At these visits, they will have a physical exam and blood tests. If they cannot visit the Clinical Center, they will be contacted by phone or have a telehealth visit.

Participation will last for about two months

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) is the disease caused by Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2). SARS-CoV-2 primarily infects the upper and lower respiratory tract and can lead to acute respiratory distress syndrome (ARDS) in a subset of patients with a known high mortality rate. Additionally, some patients develop other organ dysfunction including myocardial injury, acute kidney injury, shock along with endothelial dysfunction and subsequently micro and macrovascular thrombosis.

Much of the underlying pathology of SARS-CoV-2 is thought to be secondary to a dysregulated immune response and more recently a hypercoagulable state leading to immunothrombosis. Currently, two therapies have shown efficacy in large multicenter trials for the treatment of COVID-19, one of which is an antiviral (remdesivir) and the other is an immunosuppressant corticosteroid meant to dampen the immune response (dexamethasone).

Spleen tyrosine kinase (SYK) is a cytoplasmic tyrosine kinase involved in the intracellular signaling pathways of many different immune cells. In this pilot study we propose to use fostamatinib (an SYK inhibitor) as a targeted therapy for the immunological complications of hospitalized patients with COVID-19. The biological mechanisms by which SYK inhibition may improve outcomes in patients with COVID-19 include the inhibition of pro-inflammatory cytokines by monocytes and macrophages, decreased production of neutrophil extracellular traps (NETs) by neutrophils, and inhibition of platelet aggregation; three pathways that are mediated through Fc receptors (FcR) recognition of antigen-antibody complexes or activation of c-type lectin receptors (CLEC).

This is a randomized, double-blind, placebo-controlled trial of fostamatinib for the treatment of hospitalized patients with COVID-19.

We will randomly assign fostamatinib or matched placebo (1:1) to 60 eligible COVID-19 patients who are a 5 to 7 on the 8-point scale (requiring supplemental oxygen via nasal canula or noninvasive ventilation, requiring mechanical ventilation or extracorporeal membrane oxygenation).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patient must be hospitalized, or had their inpatient stay extended, for COVID-19.
  2. Age >=18 years
  3. Subject (or legally authorized representative) provides informed consent prior to initiation of any study procedures.
  4. Subject (or legally authorized representative) understands and agrees to comply with planned study procedures.
  5. Females of childbearing potential must agree to be abstinent or use a medical acceptable form of contraception from the time of enrollment through 30 days after last day of study drug
  6. Laboratory confirmed SARS-CoV-2 RT-PCR test within 7 days of enrollment
  7. Illness of any duration with SpO2 of less than 94% on room air requiring supplemental oxygen via nasal canula or non-invasive mechanical ventilation, or mechanical ventilation or ECMO (5 to 7 on the 8-point scale)

EXCLUSION CRITERIA:

1. ALT or AST > 5 times the upper limit of normal (ULN) or ALT or AST >= 3 x ULN and total bilirubin > 2 x ULN.
2. Estimated glomerular filtration rate (eGFR) <30ml/min
3. Pregnancy or breast feeding
4. Anticipated discharge in the next 72 hours
5. Allergy to study medication
6. Uncontrolled hypertension (systolic blood pressure >160mmHg or diastolic blood pressure >100mmHg)
7. Shock or hypotension at the time of enrollment
8. Neutrophil count <1000/microliter
9. Concern for bacterial or fungal sepsis
10. Received immunomodulatory treatment within 30 days prior to enrollment e.g., Bruton's tyrosine kinase/phosphoinositide 3 kinase/Janus kinase inhibitor or cytokine-targeting biologic therapy (anti-TNF, IL-6)
11. Received a live vaccine the last 4 weeks
12. Those who were cognitively impaired or mentally disabled prior to COVID diagnosis
13. Participation in another clinical trial for the treatment of COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Strich, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - INOVA Health Systems, Falls Church, Virginia

REFERENCES:
- [Derived] Strich JR, Tian X, Samour M, King CS, Shlobin O, Reger R, Cohen J, Ahmad K, Brown AW, Khangoora V, Aryal S, Migdady Y, Kyte JJ, Joo J, Hays R, Collins AC, Battle E, Valdez J, Rivero J, Kim IH, Erb-Alvarez J, Shalhoub R, Chakraborty M, Wong S, Colton B, Ramos-Benitez MJ, Warner S, Chertow DS, Olivier KN, Aue G, Davey RT, Suffredini AF, Childs RW, Nathan SD. Fostamatinib for the Treatment of Hospitalized Adults With Coronavirus Disease 2019: A Randomized Trial. Clin Infect Dis. 2022 Aug 24;75(1):e491-e498. doi: 10.1093/cid/ciab732. PMID 34467402
- [Derived] Strich JR, Ramos-Benitez MJ, Randazzo D, Stein SR, Babyak A, Davey RT, Suffredini AF, Childs RW, Chertow DS. Fostamatinib Inhibits Neutrophils Extracellular Traps Induced by COVID-19 Patient Plasma: A Potential Therapeutic. J Infect Dis. 2021 Mar 29;223(6):981-984. doi: 10.1093/infdis/jiaa789. PMID 33367731
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000110-H.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from October 8, 2020, through March 2, 2021 across 2 centers: Inova Fairfax Hospital (Falls Church, VA) and the National Institutes of Health (NIH) Clinical Center (Bethesda, MD).
Groups:
- Fostamatinib With Standard of Care for Treatment of COVID-19: Fostamatinib, will be administered orally at a dose of 150 mg twice daily for 14 days or 28 doses.
- Placebo With Standard of Care for Treatment of COVID-19: Placebo tablets to match fostamatinib 150 mg will be provided and administered orally at a dose of 150 mg twice daily for 14 days or 28 doses.
Period: Overall Study
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Started | 30 | 29
Completed | 27 | 24
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Death | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19 | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (13.5) | 57.0 (14.1) | 55.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 22 | 25 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 17 | 35
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 12 | 11 | 23
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59
Score on Ordinal Scale [Count of Participants; unit: Participants] — The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities.
  Participants
    Requiring supplemental oxygen | 11 | 12 | 23
    Noninvasive ventilation or high-flow oxygen devices | 17 | 15 | 32
    Invasive mechanical ventilation or extracorporeal membrane oxygen | 2 | 2 | 4
Medication for COVID-19 other than the study drug [Number; unit: participants]
  Remdesivir | 30 | 29 | 59
  Dexamethasone or other steroids (methylprednisolone and prednisone) | 30 | 29 | 59
  Convalescent plasma or monoclonal antibodies | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 1 Serious Adverse Event
Description: Number of participants with at least 1 serious adverse event by day 29 using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE is a list of common adverse event (AE) terms. Each AE term is defined and accompanied by a grading scale (1 to 5) that indicates the severity of the AE. Grading ranges from Grade 1 which is mild to Grade 5 which is death.
Time Frame: Day 29
Population: Intention-to-treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 30 | 29
Participants | 3 | 6

2. Secondary Outcome: Number of Participants With Sustained Recoveries Defined by Ordinal Scale Score of 3 or Less
Description: Time to sustained recovery determined by ordinal scale score of 3 or less and defined as time to recovery [either discharge from the hospital or hospitalization for infection control reasons only], with the recovery status sustained through day 29.
  The ordinal scale is an assessment of the clinical status. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities.
Time Frame: day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 30 | 29
Participants | 27 | 22

3. Secondary Outcome: Number of Participants Who Progress to Mechanical Ventilation
Description: Number of participants who progress to mechanical ventilation by day 29
Time Frame: day 29
Population: Participants who were not receiving mechanical ventilation at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 28 | 27
Participants | 1 | 2

4. Secondary Outcome: Number of Participants With Cumulative Clinical Endpoint of Death
Description: Number of Participants with Cumulative Clinical Endpoint of Death at Day 14, Day 28 and Day 60
Time Frame: day 14, day 28, day 60
Population: Intention-to-treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 30 | 29
Participants
  day 14 | 0 | 1
  day 28 | 0 | 3
  day 60 | 1 | 3

5. Secondary Outcome: Number of Grade 3 and 4 Adverse Events Through Day 60
Description: Number of Grade 3 and 4 AE through day 60 using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. CTCAE is a list of common adverse event (AE) terms. Each AE term is defined and accompanied by a grading scale (1 to 5) that indicates the severity of the AE. Grading ranges from Grade 1 which is mild to Grade 5 which is death.
Time Frame: Day 60
Population: Intention-to-treat analysis
Measure: Number; unit: Adverse Events
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 30 | 29
Adverse Events
  Grade 3 | 17 | 23
  Grade 4 | 3 | 7

6. Secondary Outcome: Participant Score on Ordinal Scale
Description: Participant score on ordinal scale at day 15 and day 29. The ordinal scale is an assessment of the clinical status. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities.
Time Frame: Day 15, Day 29
Population: intent to treat analysis
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Placebo With Standard of Care for Treatment of COVID-19: Placebo: Placebo tablets to match fostamatinib 150 mg will be provided and administered orally at a dose of 150 mg twice daily for 14 days or 28 doses.
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 30 | 29
score on a scale
  Day 15 | 1 [1 to 2] | 2 [1 to 5]
  Day 29 | 1 [1 to 2] | 1 [1 to 2]

7. Secondary Outcome: Change in C-Reactive Protein Levels From Baseline
Description: Change in C-Reactive Protein (CRP) blood levels from baseline. The upper limit of normal is 5 mg/L (milligrams per liter).
Time Frame: Day 3, Day 5, Day 8, Day 11, Day 15, Day 29
Population: Intent to treat analysis. 58 patients (29 in each group) provided research samples for at least one time-point since baseline except for one patient who did not take any study drug and withdrew consent after enrollment.
Measure: Median (Inter-Quartile Range); unit: mg/L (milligrams per liter)
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 29 | 29
mg/L (milligrams per liter)
  Day 3 | -37 [-94 to -6] | -46 [-105 to -1]
  Day 5 | -34 [-84 to 5] | -51 [-128 to -23]
  Day 8 | -56 [-108 to -17] | -66 [-118 to -39]
  Day 11 | -52 [-114 to -29] | -68 [-139 to -46]
  Day 15 | -43 [-109 to -33] | -71 [-126 to -47]
  Day 29 | -65 [-117 to -33] | -106 [-155 to -57]

8. Secondary Outcome: Change in Fibrinogen Levels From Baseline.
Description: Change in Fibrinogen blood levels from baseline. The upper limit of normal is Fibrinogen 466 milligrams per decilitre (mg/dL).
Time Frame: Day 3, Day 5, Day 8, Day 11, Day 15, Day 29
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: mg/dL (milligrams per decilitre)
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 29 | 29
mg/dL (milligrams per decilitre)
  Day 3 | -60 [-177 to -11] | -65 [-155 to 41]
  Day 5 | -86 [-187 to 2] | -78 [-245 to 36]
  Day 8 | -130 [-260 to -34] | -96 [-236 to -40]
  Day 11 | -141 [-277 to -77] | -138 [-250 to -14]
  Day 15 | -132 [-182 to -24] | -76 [-214 to 10]
  Day 29 | -113 [-235 to -63] | -231 [-351 to -64]

9. Secondary Outcome: Change in D-Dimer Levels From Baseline
Description: Change in D-Dimer blood levels from baseline. The upper limit of normal is 0.50 mcg/mL (microgram per milliliter).
Time Frame: Day 3, Day 5, Day 8, Day 11, Day 15, Day 29
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: mcg/mL (microgram per milliliter)
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 29 | 29
mcg/mL (microgram per milliliter)
  Day 3 | -0.01 [-0.19 to 0.25] | -0.08 [-0.4 to 0.31]
  Day 5 | -0.06 [-0.24 to 0.11] | -0.1 [-0.74 to 0.15]
  Day 8 | -0.15 [-0.74 to 0.07] | -0.24 [-1.25 to 0.1]
  Day 11 | -0.11 [-0.56 to 0.12] | -0.43 [-0.99 to 0.06]
  Day 15 | -0.06 [-0.2 to 0.12] | -0.32 [-1.02 to 0]
  Day 29 | -0.15 [-0.31 to 0] | -0.16 [-0.82 to 0.46]

10. Secondary Outcome: Change in Ferritin Levels From Baseline
Description: Change in Ferritin levels from baseline. The upper limit of normal for Ferritin is 400 mcg/L (micrograms per liter).
Time Frame: Day 3, Day 5, Day 8, Day 11, Day 15, Day 29
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: mcg/L (micrograms per liter)
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 29 | 29
mcg/L (micrograms per liter)
  Day 3 | -94 [-306 to 20] | -190 [-622 to -102]
  Day 5 | -213 [-532 to -25] | -199 [-684 to 16]
  Day 8 | -73 [-428 to 438] | -253 [-586 to -17]
  Day 11 | -169 [-853 to 93] | -491 [-756 to -239]
  Day 15 | -346 [-904 to 4] | -561 [-882 to -350]
  D29 | -578 [-1038 to -206] | -738 [-1562 to -530]

11. Secondary Outcome: Change in Interleukin 6 (IL6) Levels From Baseline
Description: Change in Interleukin 6 (IL6) blood levels from baseline. The upper limit of normal for IL6 is 1.8 picograms per milliliter (pg/mL).
Time Frame: Day 3, Day 5, Day 8, Day 11, Day 15, Day 29
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: pg/mL (picograms per milliliter)
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 29 | 29
pg/mL (picograms per milliliter)
  Day 3 | -0.7 [-11.5 to 1.4] | 1.4 [-2.6 to 6.9]
  Day 5 | -1 [-16.1 to 4.4] | 0.3 [-1.8 to 4.5]
  Day 8 | 0 [-5.5 to 3.8] | -2.5 [-6.6 to 0]
  Day 11 | -0.1 [-9.9 to 1.4] | -0.3 [-8.2 to 0.3]
  Day 15 | -1.5 [-5.5 to 1] | -0.7 [-4.3 to 0.5]
  Day 29 | -1.4 [-6.5 to -0.4] | -1.4 [-4 to -0.8]

12. Secondary Outcome: Median Days Participants Were Admitted to Intensive Care Unit
Description: Median days participants were admitted to Intensive Care Unit (ICU) by day 29
Time Frame: Day 29
Population: Participants admitted to Intensive Care Unit
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 13 | 12
Days | 3 [2 to 5] | 7 [2 to 10]

13. Secondary Outcome: Relative Change in SpO2/FiO2 Ratio
Description: Relative change in PaO2/FiO2 or SpO2/FiO2 ratio.
Time Frame: Day 3, Day 5, Day 8, Day 11, Day 15, Day 29
Population: Only SpO2/FiO2 ratio is available as PaO2 was not consistently measured. Intent to treat analysis. 58 patients (29 in each group) provided research samples for at least one time-point since baseline except for one patient who did not take any study drug and withdrew consent after enrollment.
Measure: Median (Inter-Quartile Range); unit: SpO2/FiO2 ratio
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 29 | 29
SpO2/FiO2 ratio
  Day 3 | 0.87 [0.7 to 0.97] | 0.93 [0.65 to 1.04]
  Day 5 | 1.09 [0.75 to 1.33] | 0.88 [0.76 to 1.08]
  Day 8 | 0.75 [0.59 to 1.83] | 1.09 [0.59 to 1.39]
  Day 11 | 1.49 [0.81 to 2.14] | 0.99 [0.53 to 1.59]
  Day 15 | 1.23 [0.87 to 1.5] | 1.07 [0.67 to 1.79]
  Day 29 | 0.74 [0.74 to 0.74] | 0.49 [0.42 to 0.97]

14. Secondary Outcome: Change in SOFA Score From Baseline
Description: Change in SOFA score from baseline (day 1). The Sequential Organ Failure Assessment (SOFA) Score is a mortality prediction score that is based on the degree of dysfunction of six organ systems. The score is calculated on admission and every 24 hours until discharge using the worst parameters measured during the prior 24 hours. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure). The "worst" measurement was defined as the measure that correlated to the highest number of points. The SOFA score ranges from 0 to 24.
Time Frame: Day 3, Day 5, Day 8, Day 11, Day 15, Day 29
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: score on a SOFA scale
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 29 | 29
score on a SOFA scale
  Day 3 | 0 [0 to 0] | 0 [-1 to 0]
  Day 5 | 0 [-1 to 0] | 0 [0 to 0]
  Day 8 | 0 [-1 to 1] | 0 [-1 to 0]
  Day 11 | 0 [-1 to 0] | 0 [0 to 2]
  Day 15 | -1 [-2 to 0] | 0 [-1 to 2]
  Day 29 | 0 [0 to 0] | 1 [0 to 2]

15. Secondary Outcome: Median Days on Participants Received Supplemental Oxygen
Description: Median days on participants received supplemental oxygen through day 29
Time Frame: day 29
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 30 | 29
days | 8 [5 to 10] | 20 [14 to 27]

16. Secondary Outcome: The Number of Participants That Experienced Acute Renal Failure
Description: The number of participants that experienced acute renal failure by day 29.
  Acute renal failure defined as increase in serum creatinine by ≥0.3mg/dL within 48 hours or increase in serum creatinine by ≥1.5 times baseline which is known or presumed to have occurred within the prior seven days.
Time Frame: day 29
Population: Intent to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 30 | 29
Participants | 3 | 5

17. Secondary Outcome: Number of Participants That Experienced a Deep Vein Thrombosis (DVT) or Pulmonary Embolism (PE)
Description: Number of participants that experienced a deep vein thrombosis (DVT) or pulmonary embolism (PE) by day 29
Time Frame: day 29
Population: Intent to Treat Analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 30 | 29
Participants | 2 | 0

18. Secondary Outcome: Change in Absolute Lymphocyte Count Levels From Baseline
Description: Change in Absolute lymphocyte count blood levels from baseline.
Time Frame: Day 3, Day 5, Day 8, Day 11, Day 15, Day 29
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: thousand cells per microliter
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 29 | 29
thousand cells per microliter
  Day 3 | 0.43 [0.02 to 0.64] | 0.13 [-0.18 to 0.42]
  Day 5 | 0.48 [0.08 to 1.03] | 0.38 [-0.14 to 0.73]
  Day 8 | 0.41 [0.06 to 1.22] | 0.34 [-0.02 to 1.09]
  Day 11 | 1.03 [0.15 to 1.37] | 1.02 [0.57 to 1.44]
  Day 15 | 1.03 [0.52 to 1.18] | 0.68 [0.25 to 1.07]
  Day 29 | 0.56 [0.42 to 0.89] | 0.81 [0.42 to 1.38]

19. Secondary Outcome: Change in Absolute Neutrophil Count Levels From Baseline
Description: Change in Absolute neutrophil count blood levels from baseline.
Time Frame: Day 3, Day 5, Day 8, Day 11, Day 15, Day 29
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: thousand cells per microliter
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 29 | 29
thousand cells per microliter
  Day 3 | 0.04 [-1.22 to 1.06] | -0.09 [-2.06 to 1.88]
  Day 5 | 1.53 [-2.31 to 2.5] | 0.94 [-0.97 to 2.1]
  Day 8 | 0.63 [-3.4 to 3.78] | 2.74 [-0.4 to 6.26]
  Day 11 | -0.95 [-2.34 to 1.1] | 0.85 [-1.42 to 2.6]
  Day 15 | -1.77 [-3.41 to -0.6] | -1.6 [-5.22 to 1.61]
  Day 29 | -2.54 [-4.62 to -1.12] | -2.89 [-7.9 to -0.22]

20. Secondary Outcome: Change in Platelet Count Levels From Baseline
Description: Change in Platelet count blood levels from baseline.
Time Frame: Day 3, Day 5, Day 8, Day 11, Day 15, Day 29
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: thousand cells per microliter
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
Number analyzed (Participants) | 29 | 29
thousand cells per microliter
  Day 3 | 59 [19 to 117] | 58 [24 to 103]
  Day 5 | 103 [55 to 150] | 63 [1 to 142]
  Day 8 | 145 [91 to 217] | 62 [-34 to 171]
  Day 11 | 80 [20 to 156] | 25 [-132 to 128]
  Day 15 | 11 [-30 to 92] | -26 [-198 to 26]
  Day 29 | -29 [-87 to 42] | -7 [-102 to 60]

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Fostamatinib With Standard of Care for Treatment of COVID-19 | Placebo With Standard of Care for Treatment of COVID-19
All-Cause Mortality (participants affected / at risk) | 1/30 | 3/29
Serious Adverse Events (participants affected / at risk) | 5/30 | 10/29
Other Adverse Events (participants affected / at risk) | 8/30 | 15/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostamatinib With Standard of Care for Treatment of COVID-19 (N=30) | Placebo With Standard of Care for Treatment of COVID-19 (N=29)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0
Bleeding (Gastrointestinal disorders) | 1 (1) | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Self-Extubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Post COVID Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostamatinib With Standard of Care for Treatment of COVID-19 (N=30) | Placebo With Standard of Care for Treatment of COVID-19 (N=29)
Lymphocyte count decreased (Investigations) | 4 (4) | 7 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT04579393/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT04579393/ICF_000.pdf